CLINICAL TRIAL: NCT03535480
Title: Autologous Stem Cell Ovarian Transplantation to Restore Ovarian Function in Premature Ovarian Failure Patients. Pilot Study ASCOT-2
Brief Title: Autologous Bone Marrow Stem Cell Ovarian Transplantation to Restore Ovarian Function in Premature Ovarian Failure
Acronym: ASCOT-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Antonio Pellicer, Professor, Instituto de Investigacion Sanitaria La Fe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/0251
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Premature Ovarian Failure (POF)
Keywords: ovarian reserve
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF (Experimental): Only receives G-CSF subcutaneously five days for stem cell mobilization
  Interventions: Drug: G-CSF
- ASCOT (Experimental): Receives G-CSF subcutaneously five days and then plasmapheresis for hematopoietic stem cell collection and catheterism for infusion in ovarian artery
  Interventions: Drug: G-CSF; Combination Product: ASCOT

INTERVENTIONS:
Drug: G-CSF — G-CSF subcutaneously during five days
  Other Names: Granulocyte colony stimulating factor
Combination Product: ASCOT — G-CSF subcutaneously during five days, aphaeresis to hematopoietic stem cell collection and catheterism for ovarian artery infusion
  Arms: ASCOT

SUMMARY:
This study aims to recover ovarian function in POF/POI patients. With this pueprose we designed a study protocol including two arms: ASCOT arm, were patients receive the stem cell mobilization treatment with Granulocyte colony stimulating factor (G-CSF) followed by apheresis and ovarian artery catheterism to selectively infuse the stem cells into the ovary and the G-CSF arm including patients that receive the mobilization treatment but not the ovarian artery catheterism to selectively infuse the cells into the ovary.

DETAILED DESCRIPTION:
Ovarian aging appears early in life as a decline in function at 30s leading to a complete ovarian failure around 51 years of age in women. Women in modern society have delayed the age of childbearing due to socioeconomic changes and patient´s age has become the main determinant of infertility, since it is well known that both quantity and quality of the oocytes from aging patients are seriously impaired. Nevertheless, the low ovarian reserve is not only associated with age. Primary ovarian insufficiency (POI) is a cause of infertility in women, affecting 1% of the population. It is characterized by amenorrhea, hypoestrogenism, and elevated gonadotropin levels in women younger than 40 years of age. Impairment of ovarian function in POI can be mixed up with a low ovarian reserve or poor ovarian response although represent different clinical entities and patients.

Thus, interventions to recover damaged gonads in POI patients should be developed in order to enhance their reproductive potential. Clinically, bone marrow (BM) transplant in patients with POI due to chemotherapy treatment rescues ovarian functions as demonstrated by several spontaneous pregnancies. Previous research demonstrates that autologous stem cell ovarian transplantation (ASCOT) improves ovarian reserve (AMH and AFC) in 81% of women. Three of the eleven included patients achieve 5 pregnancies and 3 healthy babies have born. Response is highly variable between patients and molecular mechanisms still unknown. New approach is mandatory to elucidate them.

Results obtained in our premature ovarian failure (POF) animal model (included chemotherapy, CT ovarian injury) demonstrate that bone marrow stem cells restore ovulation by means of increasing vascularization, proliferation and diminishing apoptosis within the ovarian niche. These ovarian niche improvements promotes follicular development, increased number of antral and preovulatory follicles and corpus luteum.

POF model is ideal to demonstrate effectivity of ASCOT technique as they represent the worst possible scene. Any improvement in those patients should be significant.

Trying to be less invasive, we designed a study protocol including two arms: ASCOT arm as previously described and Granulocyte colony stimulating factor (G-CSF) arm including patients that receive the treatment but not the apheresis nor the ovarian artery catheterism to selectively infuse the cells into the ovary.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 38 years old
* Oligo/Amenorrhea at least 4 months.
* Serum FSH > 25 IU/l, AMH < 5picomols (pM)
* Standard criteria for autologous bone marrow transplantation of our hospital.

Exclusion Criteria:

* Ovarian endometriosis
* Any ovarian surgery considered as risk factor of poor reserve.
* Genetic factors associated with poor ovarian reserve (Turner syndrome, FMR1 premutations…)
* Acquired poor ovarian reserve (Chemotherapy, radiotherapy...)
* BMI ≥ 30kg/m2.
* Iodine allergy
* Kidney failure
* Severe male factor

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Antral follicle count (AFC) | 6 months
  every antral follicle is measured

SECONDARY OUTCOMES:
Time to Menses recovery | 6 months
  Spontaneous menstrual cycle restoration and its characteristics
serum follicle stimulating hormone (FSH) and estradiol | 6 months
  serum extraction for biological measurements
ovarian reserve dynamics | 6 months
  ultrasound observation of follicular development
Controlled Ovarian Hyperstimulation (COH) response | 6 months
  ovarian response to gonadotropins
pregnancy rate | 2 years
  pregnancy rate spontaneous and after COH
Number of good quality embryos | 6 months
  Morphological criteria and developmental potential
Number of participants with treatment-related adverse events | 6 months
  Secondary effects of the received interventions following hematological and gynecological medical criteria

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, Professor, Principal Investigator — IIS la Fe
Locations (1):
- Hospital Universitario y Politécnico la Fe-IIS la Fe, Valencia, Spain